CLINICAL TRIAL: NCT05783622
Title: An Open-Label, Multicenter, Phase 1/1b Study of JANX008 in Subjects With Advanced or Metastatic Solid Tumor Malignancies
Brief Title: Study of JANX008 in Subjects With Advanced or Metastatic Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janux Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EGFR-008-001
Record Dates: First submitted 2023-03-14; First posted 2023-03-24 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Non-Small Cell Lung Cancer; Renal Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck; Colorectal Carcinoma; Small Cell Lung Cancer; Pancreatic Ductal Adenocarcinoma; Triple-negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Squamous Cell Carcinoma of Head and Neck; Colorectal Neoplasms; Small Cell Lung Carcinoma; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation (Experimental): Subjects will be dosed weekly during each 21-day cycle. Dosage per cohort will increase to determine the maximum tolerable dose.
  Interventions: Drug: JANX008
- Backfill Expansion (Experimental): Subjects will be dosed weekly during each 21-day cycle. Subjects will be dosed at levels previously declared tolerable.
  Interventions: Drug: JANX008
- Expansion (Experimental): Subjects will be dosed weekly during each 21-day cycle. Subjects will be dosed at the preliminary recommended Phase 2 dose (RP2D).
  Interventions: Drug: JANX008

INTERVENTIONS:
Drug: JANX008 — JANX008 is dosed via IV weekly in a 21-day cycle

SUMMARY:
This study is a first-in-human (FIH), Phase 1/1b, open-label, multicenter dose escalation and dose expansion study to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary anti-tumor activity of JANX008 in adult subjects with advanced or metastatic carcinoma expressing EGFR.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥18 years of age at the time of signing informed consent
* Histologically or cytologically documented locally advanced or metastatic NSCLC, SCCHN, CRC, RCC, SCLC, PDAC, TNBC
* Progressed or was intolerant to all available therapies known to confer clinical benefit appropriate for the tumor type
* Adequate organ function
* At least 1 measurable lesion per RECIST 1.1

Exclusion Criteria:

* Treatment with anti-cancer therapy within 28 days or ≤5 elimination half-lives, whichever is earlier, before enrollment
* Prior treatment with EGFR-targeted bispecific T cell engager or CAR-T cell therapy
* Prior treatment with CD3 engaging bispecific antibodies
* Clinically significant cardiovascular diseases
* Active clinically significant infection (bacterial, viral, fungal, mycobacteria, or other)
* On supplemental oxygen
* Any medical condition or clinical laboratory abnormality likely to interfere with assessment of safety or efficacy of study treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | 21 days
Incidence of Adverse Events (AE) and Serious Adverse Events (SAE) | Up to 4 years
Incidence of Clinically Significant Laboratory Abnormalities | Up to 4 years

SECONDARY OUTCOMES:
Area under the concentration time curve from time 0 to last timepoint prior to next dose JANX008 (AUC last) | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 4, 8, 9, 15, 16, 18 up to end of treatment (Up to 4 years)
Maximum observed concentration of JANX008 (Cmax) | Pre-dose and at multiple timepoints post-dose on Days 1, 2, 4, 8, 9, 15, 16, 18 up to end of treatment (Up to 4 years)
Number of participants who develop anti-drug antibodies against JANX008 | Up to 4 years
Overall Response Rate | Up to 4 years
  Proportion of participants who achieve a complete response or partial response per RECIST v1.1
Duration of Response | Up to 4 years
  Time from documentation of CR or PR to disease progression per RECIST v1.1
Progression Free Survival | Up to 4 years
  Time from treatment initiation to disease progression per RECIST v1.1
Correlation of EGFR expression level with anti-tumor activity and safety | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Janux Therapeutics, MD, Study Director — Janux Therapeutics
Locations (18):
- United States (18):
  - City of Hope Medical Center, Duarte, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - University of California San Diego Moores Cancer Center, San Diego, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center NYU Langone Health, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas